CLINICAL TRIAL: NCT03728920
Title: Screening Muscle Strength in Arthroscopic Surgery of the Hip
Acronym: SMASH
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Arman Memarzadeh, Clinical and Research Fellow, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: SMASH V9
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Femoroacetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Muscle strength measurement — Patients awaiting hip arthroscopy will undergo muscle strength testing pre- and post-operatively. There will be no deviation of treatment from their NHS care. Validated outcome measure questionnaires will be completed at five months post-operatively. Magnetic resonance imaging and electromyography tests will be performed on a subset of patients post-operatively.

SUMMARY:
Hypothesis We hypothesise that hip muscle strength can predict the outcome of hip arthroscopy. A relationship between strength and outcome can improve the success of the procedure and avoid unnecessary and potentially harmful surgery.

Objectives The primary objective is to evaluate the relationship between hip muscle strength and outcomes of hip arthroscopy. The secondary objective is to determine a 'threshold strength' above which the operation becomes successful. If this relationship is established, it would launching a randomised control trial with targeted physiotherapy as the intervention.

Background Hip arthroscopy is key-hole surgery to the hip joint which is performed for femoroacetabular impingement; a condition which describes a shape mismatch between the ball-and-socket hip joint. The number of procedures is increasing, however, studies have shown success in only half of patients undergoing the procedure.

Several factors have been linked with outcomes; however, the influence of muscle strength has never been investigated. We performed a systematic review of this topic, revealing that muscles around affected hips are significantly weaker. We also developed a standardised protocol for the measurement of muscle strength.

Plan Patients awaiting hip arthroscopy will undergo muscle strength testing pre- and post-operatively. There will be no deviation of treatment from their NHS care. Validated outcome measure questionnaires will be completed at five months post-operatively. Magnetic resonance imaging and electromyography tests will be performed on a subset of patients post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-45 years with evidence of FAI on MRI scan (the standard method of imaging of the condition in the NHS)
* Competent to consent to study participation

Exclusion Criteria:

* Established osteoarthritis with evidence of osteophytes (Tonnis grade >2)
* Patient with hip dysplasia (centre-edge-angle <20 degrees)
* Patients with full thickness cartilage (chondral) lesions
* Previous diagnosis of mental health disorder
* Failure to comply with Addenbrooke's hospital post-operative rehabilitation exercises tailored to hip arthroscopy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young adult patients suffering with femoroacetabular impingement, prior to the development of arthritis
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-01-10 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Hip Outcome Score | 6 months post-operatively
  Patient reported outcome measure to assess the success of hip arthroscopy

IPD SHARING:
Plan to Share IPD: No